CLINICAL TRIAL: NCT05600842
Title: De-escalated Radiation for Human Papillomavirus-Positive Squamous Cell Carcinoma of the Oropharynx
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Eric Chen, Assistant Professor, University of California, Irvine
Other Study IDs: 2048; UCI 22-132 (Other: CFCCC)
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- De-escalated radiotherapy
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — IMRT will be given in 30 daily fractions at 2 Gy per fraction (60 Gy total) beginning Day 1; Six fractions will be delivered per week. High risk patients will receive induction chemotherapy with 2 cycles of carboplatin and paclitaxel.

SUMMARY:
This is a single-arm, observational registry study determining the effects of reduced radiation dose in select patients with human papillomavirus (HPV) positive oropharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven (from primary lesion and/or lymph nodes) diagnosis of human papillomavirus (HPV)-positive oropharyngeal squamous cell carcinoma. HPV-positivity will be defined as tumors that are p16-positive by immunohistochemistry. Numerous studies have demonstrated near 100% agreement between p16 and HPV for patients with oropharyngeal cancer. As such, the use of p16 has been accepted as an appropriate surrogate for HPV status.
* Clinical stage I, II, or III disease (AJCC Eighth Edition); Note: Patients with M1 tumors (distant metastases) are not eligible;
* History/physical examination within 6 weeks prior to registration, including assessment of weight and recent weight loss;
* Age ≥ 18;
* PET/CT within 6 weeks prior to registration;
* Patients must sign a study-specific informed consent form prior to study entry.
* Both men and women and members of all races and ethnic groups are eligible for this trial. Non-English speaking, deaf, hard of hearing and illiterate individuals are eligible for this trial.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years;
* Patients who have had initial surgical treatment other than the diagnostic biopsy of the primary site or nodal sampling of the neck disease are excluded;
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
* Receipt of prior radiotherapy that would result in overlap with proposed field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HPV-positive oropharyngeal cancer
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
2-Year Progression-Free Survival | Given the natural history of this disease, PFS will be monitored up to 2 years from registration
  Progression-free survival (PFS) is defined as the time from registration to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival | Given the natural history of this disease, overall survival will be monitored for up to 2 years from registration
  Survival time will be measured from the date of randomization to the date of death due to any cause or last follow-up.
Local-regional control | Given the natural history of this disease, local-regional control will be monitored up to 2 years from registration
  Local-regional control is defined as the absence of local and/or regional progression.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No